CLINICAL TRIAL: NCT00315731
Title: A Multi-Center Study to Examine the Pharmacokinetics, Whole Body and Organ Dosimetry, and Biodistribution of Fission-Derived Iodine I 131 Tositumomab for Patients With Previously Untreated or Relapsed Follicular or Transformed Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study Of Pharmacokinetics, Whole Body And Organ Dosimetry, And Biodistribution Of Fission-Derived Iodine I 131 Tositumomab (BEXXAR®) For Patients With Previously Untreated Or Relapsed Follicular Or Transformed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/027
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma, Follicular
Keywords: Bexxar; tositumomab and iodine I 131 tositumomab therapeutic regiment; fission; Non-Hodgkin's lymphoma; Iodine I 131 Tositumomab; pharmacokinetics; tellurium
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin

ARMS (1):
- tositumomab and iodine I 131 tositumomab (Experimental): Subjects participating in this study will receive a standard 5 mCi dosimetric dose of fission-derived Iodine I-131 tositumomab, immediately following an infusion of 450 mg of unlabeled tositumomab. Using the dosimetric data from three of the six imaging time points and the subject's weight, a patient-specific activity (mCi) of Iodine I-131 will be calculated to deliver the desired total body dose of radiation (75 cGy). All subjects will then receive an infusion of unlabeled tositumomab (450 mg) immediately followed by an infusion of the subject specific dose of tellurium-derived Iodine I-131 tositumomab (35 mg) to deliver a total body dose (TBD) of 75 cGy.
  Interventions: Biological: Follicular Lymphoma

INTERVENTIONS:
Biological: Follicular Lymphoma — For subjects with previously untreated or relapsed follicular or transformed follicular non-Hodgkin's

SUMMARY:
Patients will receive a standard 5 mCi dosimetric dose of fission-derived Iodine I 131 Tositumomab. Pharmacokinetic data for the primary endpoint analysis will be derived from testing done on blood samples drawn at 12 timepoints over the first 7 days following administration of the dosimetric dose. Whole body gamma camera images will be obtained on six days following the dosimetric dose. Organ and tumor dosimetry data will be generated from gamma camera counts of specific organs and tumor. All scans will be examined by an independent review panel to evaluate biodistribution of the radionuclide.

Using the dosimetric data from three of the six imaging time points and the patient's weight, a patient-specific activity (mCi) of Iodine-131 will be calculated to deliver the desired total body dose of radiation (75 cGy). Patients will receive an infusion of unlabeled Tositumomab (450 mg) immediately followed by an infusion of the patient specific dose of tellurium-derived Iodine I 131 Tositumomab (35 mg) to deliver a total body dose (TBD) of 75 cGy. Patients will be followed closely obtaining safety information during the post-treatment period, and for response and safety at 3,6,and 12 months during the first year, annually thereafter up to five years, and annually for additional safety and outcomes information up to 10 years.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years of age
2. A histologically confirmed diagnosis of the following:

   Follicular lymphoma, Grade 1, 2, or 3 or diffuse large cell lymphoma concurrent with or following the diagnosis of follicular lymphoma (World Health Organization/Revised European-American Lymphoma [WHO/REAL] classification).

   International Working Formulation histological equivalents included:

   Follicular, small-cleaved; Follicular, mixed small-cleaved and large-cell; Follicular large-cell; or Transformed diffuse large-cell lymphoma following or concurrent with a diagnosis of follicular lymphoma.
3. Stage III or IV disease at the time of study entry (based on Ann Arbor Staging Classification)
4. Previously untreated or recurrent lymphoma after no more than 4 prior qualifying therapy regimens; steroids alone, as treatment for lymphoma, not considered a treatment regimen
5. Performance status of at least 70% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
6. Bi dimensionally measurable disease with at least one lesion measuring greater than or equal to 2.0 cm x 2.0 cm (greater than or equal to 4.0 cm2) by computed tomography (CT) scan
7. Absolute B lymphocyte count (as determined by CD19 reactivity [flow cytometric determination of CD19+ B lymphocyte count]) of 30 to 350 cell/mm3 within 21 days prior to study enrollment
8. Absolute neutrophil count greater than or equal to 1500 cells/mm3; platelet count greater than or equal to 150,000/mm3; and hemoglobin greater than or equal to 10 g/dL within 21 days prior to study enrollment; blood products and/or growth factors not taken within 4 weeks prior to blood draw
9. Adequate renal function, defined as serum creatinine <1.5 x upper limit of normal (ULN), and hepatic function, defined as total bilirubin <1.5 x ULN and aspartate transaminase (AST) <5 x ULN, within 21 days of study enrollment
10. HAMA negative within 21 days prior to study enrollment
11. Signed IRB approved consent form prior to any study-specific procedures being implemented

Exclusion criteria

1. Greater than 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 90 days of study enrollment; a unilateral bone marrow biopsy was adequate; marrow core was greater than or equal to 2.0 cm in length
2. Prior chemotherapy, biologic therapy, steroids, or radiation therapy as treatment for NHL within 28 days prior to study enrollment; subjects receiving low doses of steroids for non neoplastic disease acceptable to enter this study ("Low dose steroids" was defined as less than or equal to 10 mg of prednisone or equivalent per day.)
3. Prior rituximab therapy within 120 days prior to study enrollment
4. Prior radioimmunotherapy
5. Prior splenectomy
6. Splenomegaly defined as spleen mass greater than 700 grams, where splenic mass was defined as follows:

   Spleen mass = л(X x Y x Z)/6 Where X and Y are the greatest perpendicular diameters in cm on any single CT scan slice, and Z is the number of CT scan slices upon which the spleen is visible times the slice thickness in cm
7. Bulky disease as defined as any uni-dimensional measurement of lymphomatous mass exceeding 7 cm
8. Prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the subject had a generally accepted risk of recurrence less than 20%
9. Central nervous system involvement by lymphoma
10. Evidence of active infection requiring IV antibiotics at the time of study enrollment
11. Known human immunodeficiency virus (HIV) infection
12. New York Heart Association Class III or IV heart disease or other serious illness that would preclude evaluation.
13. Active obstructive hydronephrosis
14. Evidence of clinically significant ascites or pleural effusion observed on screening physical examination or baseline CT scan
15. Prior myeloablative therapy
16. History of failed stem cell collection
17. Pregnant or nursing subjects (Subjects of childbearing potential had to have a negative serum pregnancy test within 21 days of study enrollment. Males and females of childbearing age had to agree to use effective contraception for up to 12 months after the radioimmunotherapy.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03-31 (Actual); Primary Completion 2006-12-04 (Actual); Study Completion 2013-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 393229/027 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/393229/027?search=study&study_ids=393229%2F027#rs
- Available data/document: Study Protocol: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 393229/027 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Blood pharmacokinetics (the primary objective), biodistribution, and organ dosimetry following a dosimetric dose of tositumomab and fission-derived iodine I-131 tositumomab in this study were compared with results following a dosimetric dose of tositumomab and tellurium-derived iodine I-131 tositumomab in a historical control group (NCT00996996).
Groups:
- Tositumomab and Fission-derived Iodine I-131 Tositumomab: Dosimetric dose (administered only once on Day 0): 450 milligrams (mg) unlabeled tositumomab administered intravenously (IV) for 1 hour, followed immediately by 5 millicurie (mCi) fission-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. Therapeutic dose (administered only once on Day 7): 450 mg unlabeled tositumomab administered IV for 1 hour, followed immediately by Tellurium-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. The dose was calculated based on the dosimetric dose results to deliver a total body radiation dose of 75 centigray (cGy).
Period: Overall Study
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Started | 15
Completed | 9
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) at 0 to 120, 0 to 168, and 0 to Infinity Hours
Description: Area under the concentration-time curve for 131I-tositumomab from time 0 to 120, 0 to 168, and time 0 to infinity hours (extrapolated), after the end of the dosimetric dose infusion. Unit: %ID.h/mL, where %ID/mL is the percentage of the injected dose per milliliter blood. AUC measures how much drug is in the system over time after infusion.
Time Frame: 0-120, 0-168, and 0-infinity hours from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID.h/mL
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
%ID.h/mL
  AUC(0-120) | 1.04 [0.88 to 1.24]
  AUC(0-168) | 1.18 [0.98 to 1.43]
  AUC(0-infinity) | 1.39 [1.10 to 1.75]

2. Primary Outcome: Maximum Concentration (Cmax) Values
Description: Cmax is the maximum observed 131I-tositumomab concentration from time zero (end of the dosimetric dose infusion) to 7 days after the end of the infusion. Unit: %ID/mL, where %ID/mL is the percentage of the injected dose per milliliter blood. Cmax is the highest drug concentration in the blood after infusion.
Time Frame: 0 to 7 days from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID/mL
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
%ID/mL | 0.0189 [0.0169 to 0.0211]

3. Primary Outcome: Terminal Phase Half-life (t½)
Description: The terminal phase half-life of 131 I tositumomab in hours. Half-life measures how long it takes for the concentration of drug in the blood to decrease by half.
Time Frame: 0 to 7 days from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
hours | 59.5 [48.8 to 72.5]

4. Primary Outcome: Clearance (CL) Values
Description: Clearance of 131I-tositumomab after intravenous administration. The clearance of a drug measures the rate at which the drug is removed from the body after the dose.
Time Frame: 0 to 7 days from dosimetric dose given only once on Day 0
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters per hour (ml/hr)
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
milliliters per hour (ml/hr) | 71.9 [57.1 to 90.6]

5. Primary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution at steady state of 131I-tositumomab. Volume of distribution measures how much the drug spreads through the body after the dose.
Time Frame: 0 to 7 days from dosimetric dose given only once on Day 0
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters (ml)
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11
milliliters (ml) | 6055 [5293 to 6927]

6. Secondary Outcome: Area Under the Curve (AUC) at 0 to 120 Hours
Description: Area under the concentration-time curve from time 0 to 120 hours after the end of the dosimetric dose infusion. Unit: %ID.h/mL, where %ID/mL is the percentage of the injected dose per milliliter blood. AUC measures how much drug is in the system over time after infusion.
Time Frame: 0-120 hours from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID.h/mL
Groups:
- Tellurium-Derived Iodine I-131 Tositumomab: Evaluable participant data from the historical trial, Study RIT II 003 (NCT01224821), in which participants received tisitumomab and tellurium-derived iodine I-131 tositumomab dosimetric dose (administered only once on Day 0): 450 milligrams (mg) unlabeled tositumomab administered intravenously (IV) for 1 hour, followed immediately by 5 millicurie (mCi) tellurium-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. Therapeutic dose (administered only once on Day 7): 450 mg unlabeled tositumomab administered IV for 1 hour, followed immediately by Tellurium-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. The dose was calculated based on the dosimetric dose results to deliver a total body radiation dose of 75 centigray (cGy).
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11 | 22
%ID.h/mL | 1.04 [0.88 to 1.24] | 1.07 [0.98 to 1.17]
Statistical Analysis 1: Comparison: Tositumomab and Fission-derived Iodine I-131 Tositumomab vs Tellurium-Derived Iodine I-131 Tositumomab; Test type: Non-Inferiority or Equivalence — Comparability of AUC values after dosimetric dose of fission-derived 131I-tositumomab with historical data from tellurium-derived 131I-tositumomab; Ratio of AUC(0-120) = 0.97, 90% CI 2-sided [0.85 to 1.12] — Ratio of AUC(0-120) is the ratio of AUC(0-120) values following infusion of fission-derived 131I-tositumomab to those following infusion of tellurium-derived 131I-tositumomab

7. Secondary Outcome: Area Under the Curve (AUC) at 0 to 168 Hours
Description: Ratio and 90% confidence interval for AUC(0-168) after dosimetric dose of fission-derived 131I-tositumomab to historical data from tellurium-derived 131I-tositumomab. AUC measures how much drug is in the blood over time after the dose.
Time Frame: 0-168 h from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID.h/mL
Groups:
- Tellurium-Derived Iodine I-131 Tositumomab: Evaluable participant data from the historical trial, Study RIT II 003 (NCT01224821), in which participants received tisitumomab and tellurium-derived iodine I-131 tositumomab Dosimetric dose (administered on Day 0): 450 milligrams (mg) unlabeled tositumomab administered intravenously (IV) for 1 hour, followed immediately by 5 millicurie (mCi) tellurium-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. Therapeutic dose (administered on Day 7): 450 mg unlabeled tositumomab administered IV for 1 hour, followed immediately by Tellurium-derived iodine I-131 tositumomab (contained in 35 mg tositumomab) administered IV for 20 minutes. The dose was calculated based on the dosimetric dose results to deliver a total body radiation dose of 75 centigray (cGy).
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11 | 22
%ID.h/mL | 1.18 [0.98 to 1.43] | 1.24 [1.13 to 1.35]
Statistical Analysis 1: Comparison: Tositumomab and Fission-derived Iodine I-131 Tositumomab vs Tellurium-Derived Iodine I-131 Tositumomab; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio of AUC(0-168) = 0.96, 90% CI 2-sided [0.83 to 1.11] — Ratio of AUC(0-168) is the ratio of AUC(0-168) values following infusion of fission-derived 131I-tositumomab to those following infusion of tellurium-derived 131I-tositumomab

8. Secondary Outcome: Area Under the Curve (AUC) at 0 to Infinity (Extrapolated)
Description: Ratio and 90% CI for AUC (0 to infinity) after dosimetric dose of fission-derived 131I-tositumomab to historical data from tellurium derived 131I-tositumomab. AUC measures how much drug is in the blood over time after the dose is given.
Time Frame: 0 to infinity h from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID.h/mL
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11 | 22
%ID.h/mL | 1.39 [1.10 to 1.75] | 1.50 [1.35 to 1.67]
Statistical Analysis 1: Comparison: Tositumomab and Fission-derived Iodine I-131 Tositumomab vs Tellurium-Derived Iodine I-131 Tositumomab; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio of AUC(0 to infinity) = 0.93, 90% CI 2-sided [0.78 to 1.10]

9. Secondary Outcome: Maximum Concentration (Cmax) Values
Description: Maximum observed concentration from time zero (end of the dosimetric dose infusion) to 7 days after the end of the infusion. Unit: %ID/mL, where %ID/mL is the percentage of the injected dose per milliliter blood. Cmax is the highest drug concentration in the blood after the dose.
Time Frame: 0 to 7 days from dosimetric dose (given only once on Day 0)
Population: All participants considered as evaluable for pharmacokinetic assessment per protocol criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: %ID/mL
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 11 | 22
%ID/mL | 0.0189 [0.0169 to 0.0211] | 0.0193 [0.0176 to 0.0211]
Statistical Analysis 1: Comparison: Tositumomab and Fission-derived Iodine I-131 Tositumomab vs Tellurium-Derived Iodine I-131 Tositumomab; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio of Cmax = 0.98, 90% CI 2-sided [0.87 to 1.11]

10. Secondary Outcome: Mean Residence Times From Day 0 to Day 7
Description: Whole body images from anterior and posterior gamma camera scans were collected to assess dosimetry. Assessment of organ dosimetry required gamma camera scans from at least 4 time points. Nuclear medicine reviewers conducted a visual examination of the gamma camera scans and calculated the total body residence times. Residence time is calculated from the rate of total body clearance of iodine I-131 radioactivity during the dosimetric dose. Residence time is a measure of how long the drug resides in the body.
Time Frame: 0 to 7 days from dosimetric dose (given only once on Day 0)
Population: All participants who were considered evaluable for dosimetric assessment per protocol eligibility criteria and had gamma camera scans from at least 4 time points. Different numbers of participants were analyzed for different organs (represented by n=X, X in the category titles).
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 10 | 22
hours
  Total Body, n=10, 22 | 87.9 [78.8 to 96.9] | 95.7 [90.8 to 100.7]
  Kidneys, n=10, 21 | 1.5 [1.2 to 1.7] | 1.9 [1.7 to 2.1]
  Liver, n=10, 22 | 3.7 [3.0 to 4.4] | 4.7 [4.2 to 5.3]
  Lungs, n=9, 22 | 3.0 [2.4 to 3.5] | 4.3 [3.8 to 4.8]
  Spleen, n=10, 22 | 1.3 [1.1 to 1.6] | 1.8 [1.5 to 2.1]
  Urinary Bladder, n=10, 22 | 1.6 [1.5 to 1.7] | 1.4 [1.3 to 1.4]
  Remainder of Body, n=10, 22 | 76.1 [66.9 to 85.4] | 81.7 [77.1 to 86.4]

11. Secondary Outcome: Mean Absorbed Dose in the Source Organs and the Target Organs
Description: The radiation absorbed dose to source organs were determined with Organ Level Internal Dose Assessment/Exponential Modeling (OLINDA/EXM) software using residence times directly determined by an independent reviewer for kidneys, liver, lungs, spleen, urinary bladder, and total body; the radiation absorbed dose for the remaining target organs was based on a mathematical model used to calculate source organ radiation dose estimates using the same OLINDA/EXM software. OLINDA/EXM is a registered proprietary computer program.
Time Frame: 0 to 7 days from dosimetric dose
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: mGy/MBq
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 10 | 22
mGy/MBq
  Total Body | 0.23 [0.20 to 0.25] | 0.25 [0.23 to 0.26]
  Adrenals | 0.25 [0.23 to 0.28] | 0.28 [0.26 to 0.29]
  Brain | 0.19 [0.17 to 0.21] | 0.2 [0.19 to 0.21]
  Breast | 0.18 [0.16 to 0.20] | 0.2 [0.19 to 0.21]
  Gallbladder Wall | 0.26 [0.23 to 0.28] | 0.28 [0.27 to 0.30]
  Heart Wall | 0.24 [0.21 to 0.26] | 0.26 [0.24 to 0.27]
  Kidneys | 0.72 [0.61 to 0.83] | 0.92 [0.83 to 1.01]
  Lower Large Intestine Wall | 0.24 [0.21 to 0.27] | 0.26 [0.24 to 0.27]
  Liver | 0.36 [0.30 to 0.41] | 0.45 [0.40 to 0.49]
  Lungs | 0.44 [0.37 to 0.52] | 0.61 [0.55 to 0.68]
  Muscle | 0.21 [0.18 to 0.23] | 0.22 [0.21 to 0.24]
  Osteogenic Cells | 0.44 [0.40 to 0.49] | 0.45 [0.42 to 0.47]
  Ovaries | 0.25 [0.22 to 0.27] | 0.26 [0.25 to 0.28]
  Pancreas | 0.26 [0.24 to 0.29] | 0.29 [0.28 to 0.31]
  Red Marrow | 0.24 [0.18 to 0.30] | 0.20 [0.19 to 0.21]
  Skin | 0.17 [0.15 to 0.19] | 0.19 [0.18 to 0.20]
  Small Intestine | 0.24 [0.22 to 0.27] | 0.26 [0.25 to 0.27]
  Spleen | 0.79 [0.50 to 1.08] | 0.84 [0.72 to 0.96]
  Stomach | 0.24 [0.21 to 0.26] | 0.26 [0.25 to 0.27]
  Testes | 0.21 [0.18 to 0.23] | 0.22 [0.21 to 0.23]
  Thymus | 0.22 [0.19 to 0.24] | 0.23 [0.22 to 0.25]
  Thyroid | 0.21 [0.19 to 0.23] | 0.25 [0.20 to 0.29]
  Upper Large Intestine Wall | 0.24 [0.21 to 0.27] | 0.26 [0.26 to 0.27]
  Urinary Bladder Wall | 0.73 [0.73 to 0.74] | 0.66 [0.66 to 0.69]
  Uterus | 0.26 [0.23 to 0.28] | 0.27 [0.27 to 0.28]

12. Secondary Outcome: Number of Participants With Expected Distribution of Radioactivity in the Circulatory System Compared With Uptake by Other Organs.
Description: Expected biodistribution (images): most radioactivity (RA) in blood pool, with uptake in normal liver and spleen less than the heart. Later time points, RA in blood pool decrease and uptake in normal liver and spleen decrease. Images may show uptake by the thyroid gland, kidneys, urinary bladder, and lungs. Altered biodistribution: Blood pool not visualized or diffuse, intense uptake in the liver and/or spleen, or uptake suggestive of urinary obstruction, diffuse lung uptake greater than the blood pool
Time Frame: 0 to 7 days from dosimetric dose (given only once on Day 0)
Population: All participants who were considered evaluable for dosimetric assessment per protocol eligibility criteria and had gamma camera scans from at least 4 time points.
Measure: Number; unit: participants
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab | Tellurium-Derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 10 | 22
participants | 10 | 22

13. Secondary Outcome: Percentage of Participants Evaluable for Confirmed Response With Complete Response (CR), CR Unconfirmed (CRu), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD)
Description: Evaluation based on the Int'l Workshop to Standardize Response Criteria for non-Hodgkin's Lymphoma (NHL). CR, complete disappearance of all detectable clinical/radiographic evidence of disease, disappearance of all disease-related symptoms if present before therapy, and normalization of biochemical abnormalities definitely assignable to NHL. CRu, complete response unconfirmed, included complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities definitely assignable to NHL. PR, >=50% decrease in sum of perpendicular diameters (SPD) of all measurable lesions determined at baseline. SD, less than a PR but not progressive disease (>=50% increase from nadir in SPD for all measurable disease or the appearance of any new lesion that was >=1.4 cm x 1.4 cm by radiographic evaluation or >=1.0 cm by palpation per physical examination).
Time Frame: From Baseline up to 99 Months
Population: ITT-E Population. The individual categories for confirmed CR, confirmed CRu, etc. counts those participants who had their response confirmed by the exact same response, not those who had their response confirmed by a better response (for example, Cru to CR; PR to CR; PR to CRU; etc.).
Measure: Number; unit: percentage of participants
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 15
percentage of participants
  Overall response (CR, CRu, or PR) | 67
  CR | 33
  PD | 7
  CRu | 7
  PR | 27
  SD | 7

14. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from first documented response (CR, CRu, or PR) until disease progression.
Time Frame: Week 7 to Week 260 post treatment
Population: ITT-E Population. Only participants who had a response (CR, CRu, or PR) were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 10
months | NA [NA to NA] — The median was not reached using Kaplan-Meier methodology because not enough events were observed.

15. Secondary Outcome: Progression-free Survival
Description: Progression-free survival, or time to progression, is defined as the time from the dosimetric dose to the first documented disease progression (PD) or death. PD is defined as a >= 50% increase from nadir in the SPPD for all measurable disease.
Time Frame: Week 7 to Week 260 post treatment
Population: ITT-E Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 15
months | 59.0 [10.1 to NA] — An upper limit of the 95% confidence interval could not be calculated due to the low number of events.

16. Secondary Outcome: Overall Survival
Description: Time to death is defined as the time from the dosimetric dose to the date of death.
Time Frame: Week 7 to Week 260 post treatment
Population: ITT-E Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Number analyzed (Participants) | 15
months | NA [NA to NA] — The median was not reached using Kaplan-Meier methodology due to the low number of events.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs occurring from the time of enrollment up to 99 months are reported.
Description: An on-therapy adverse event (AE) is an AE that occurred from the time of enrollment until 26 weeks after the dosimetric dose (DD) or until administration of subsequent therapy for lymphoma, whichever occurred first. After Week 26, AEs were reported if considered by the investigator to be possibly associated with the iodine I-131 tositumomab DD.
Arm/Group | Tositumomab and Fission-derived Iodine I-131 Tositumomab
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Fission-derived Iodine I-131 Tositumomab (N=15)
Pyrexia (General disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Fission-derived Iodine I-131 Tositumomab (N=15)
Fatigue (General disorders) | 6
Pyrexia (General disorders) | 5
Chills (General disorders) | 4
Axillary pain (General disorders) | 2
Local swelling (General disorders) | 2
Pain (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Edema peripheral (General disorders) | 1
Swelling (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Abdominal discomfort (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestions (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorhea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Hordeolum (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper resp trct infection (Infections and infestations) | 1
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/oral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypothyroidism (Endocrine disorders) | 3
Eyelid margin crusting (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Pelvic discomfort (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Dysuria (Renal and urinary disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Absolute neutrophil count (calc) <1000 cells/millimeter^3 (Investigations) | 8
White Blood Cell count <2000 cells/millimeter^3 (Investigations) | 5
Platelets <50000 cells/millimeter^3 (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.